CLINICAL TRIAL: NCT01293487
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, TOLERABILITY, IMMUNOGENICITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF ESCALATING DOSES OF RN564 IN WOMEN WITH OSTEOPENIA AND IN HEALTHY MEN
Brief Title: Safety And Tolerability Study Of RN564 In Women With Osteopenia And Healthy Men.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1151001
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-06

CONDITIONS: Osteopenia; Osteoporosis; Bone Disease
Keywords: Phase 1; Osteopenia; RN564
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Bone Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: RN564

INTERVENTIONS:
Biological: RN564 — Intravenous, single dose with experimental dose

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RN564 in women with osteopenia and healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteopenia for women (BMD T-scores between -1.0 and - 2.5 SD at the lumbar spine, the femoral neck or total hip)
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* Have at least 3 vertebral bodies in the L1-L4 region and one femoral neck site that are accessible by DXA.

Exclusion Criteria:

* Evidence or history of any underlying condition, other than primary osteopenia, that affect bone metabolism (eg, hyperparathyroidism, hypoparathyroidism).
* Subjects with pre-existing periodontal/dental disease or those who have undergone invasive dental procedures (eg, tooth extraction, oral surgery) within 60 days prior to Day -1.
* If QTcF exceeds 455 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2012-05-24 (Actual); Study Completion 2012-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Ambulatory Diagnostic Center, Coral Gables, Florida
  - Gable Diagnostics, Coral Gables, Florida
  - Gables Diagnostics, Coral Gables, Florida
  - SeaView Research, Inc., Miami, Florida
  - Miami Research Associates, Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1151001&StudyName=Safety%20And%20Tolerability%20Study%20Of%20RN564%20In%20Women%20With%20Osteopenia%20And%20Healthy%20Men.

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04840082 0.3 mg/kg: Healthy postmenopausal female participants with osteopenia between the ages of 55-80 years received a single intravenous (IV) infusion of PF-04840082 0.3 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 1.0 mg/kg: Healthy postmenopausal female participants with osteopenia between the ages of 55-80 years received a single IV infusion of PF-04840082 1.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 6.0 mg/kg: Healthy postmenopausal female participants with osteopenia between the ages of 55-80 years received a single IV infusion of PF-04840082 6.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 24.0 mg/kg: Healthy postmenopausal female participants with osteopenia between the ages of 55-80 years received a single IV infusion of PF-04840082 24.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 3.0 mg/kg: Healthy postmenopausal female participants with osteopenia and healthy male participants between the ages of 55-80 years received a single IV infusion of PF-04840082 3.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 12.0 mg/kg: Healthy postmenopausal female participants with osteopenia and healthy male participants between the ages of 55-80 years received a single IV infusion of PF-04840082 12.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- PF-04840082 18.0 mg/kg: Healthy postmenopausal female participants with osteopenia and healthy male participants between the ages of 55-80 years received a single IV infusion of PF-04840082 18.0 mg/kg over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
- Placebo: Healthy postmenopausal female participants with osteopenia and healthy male participants between the ages of 55-80 years received a single IV infusion of matching placebo over 60 minutes on Day 1 following an overnight fast of at least 6 hours.
Period: Overall Study
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
Completed | 6 | 6 | 6 | 5 | 8 | 8 | 8 | 18
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (6.3) | 65.0 (9.8) | 61.0 (4.2) | 63.3 (5.2) | 61.3 (5.5) | 63.6 (7.2) | 61.3 (5.2) | 62.8 (5.1) | 62.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 4 | 4 | 4 | 14 | 50
  Male | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting or Intolerable Treatment Related Adverse Events (AEs)
Description: Dose-limiting or intolerable treatment related AEs was defined as any of the following criteria occurred in 2 or more participants: Serious adverse events, Increased liver transaminases, Increased bilirubin (in absence of ALT/AST elevations, allergic / hypersensitivity reactions, vasculitis, Musculoskeletal pain, Increased serum creatinine, Diarrhea, enteritis or nausea, Prolongation of QTcF interval or any other criteria If considered appropriate by the Medical Monitor and Investigator. A dose level was also be considered intolerable if, in the judgment of the Investigator and Sponsor, the type, frequency, or severity of AEs becomes unacceptable.
Time Frame: Day 1 to Day 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With All-Causality AEs by Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: Day 1 to Day 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage of participants
  Grade 1 | 100.0 | 50.0 | 100.0 | 66.7 | 62.5 | 37.5 | 62.5 | 60.0
  Grade 2 | 0 | 16.7 | 0 | 16.7 | 0 | 25.0 | 12.5 | 10.0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing/Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Treatment-Related AEs by Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Relatedness to drug was assessed by investigator.
Time Frame: Day 1 to Day 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage of participants
  Grade 1 | 50.0 | 16.7 | 50.0 | 33.3 | 50.0 | 0 | 37.5 | 20.0
  Grade 2 | 0 | 16.7 | 0 | 0 | 0 | 12.5 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing/Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Any Laboratory Abnormality
Description: Criteria for abnormality: hematology: hemoglobin, hematocrit, red blood cell count: less than(<) 0.8*lower limit of normal (LLN); platelets: <0.5*LLN,>1.75*ULN, white blood cell count: <0.6*LLN, >1.5*ULN; lymphocytes, total neutrophils: <0.8*LLN, >1.2*ULN; eosinophils, basophils, monocytes: >1.2*ULN; coagulation: activated partial thromboplastin time, prothrombin, prothrombin international ratio: >1.1*ULN; liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function: blood urea nitrogen, creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium>1.05*ULN, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN), urine casts, granular casts, hyaline casts>1 LPF; hormones: T4, T3, TSH<0.8*LLN.
Time Frame: Day 1 to 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
Participants | 3 | 3 | 4 | 1 | 3 | 4 | 4 | 12

5. Primary Outcome: Median Change From Baseline in Platelets and White Blood Cell [WBC] Count (With Differentials) at Last Observation
Description: Median change from baseline in platelets, WBC count, lymphocytes (absolute [Abs]), total neutrophils (Abs), basophils (Abs), eosinophils (Abs), and monocytes (Abs)
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: 10^3 cells/millimeter cube (mm^3)
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
10^3 cells/millimeter cube (mm^3)
  Platelets | 8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -9 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -31 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  White Blood Cell Count | -0.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.9 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Lymphocytes (Abs) | -0.10 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.06 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.06 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.06 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.07 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.05 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.09 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Total Neutrophils (Abs) | -0.78 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.04 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.34 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.51 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.12 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.61 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.11 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.35 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Basophils (Abs) | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Eosinophils (Abs) | 0.03 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.04 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Monocytes (Abs) | -0.10 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.04 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.04 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.03 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.03 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.00 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

6. Primary Outcome: Median Change From Baseline in Red Blood Cell (RBC) Count at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: 10^6 cells/mm^3
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
10^6 cells/mm^3 | -0.05 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.07 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.14 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.10 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.05 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.30 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.06 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.07 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

7. Primary Outcome: Median Change From Baseline in Hematocrit at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: percentage of red blood cells
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
percentage of red blood cells | 0.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -2.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

8. Primary Outcome: Median Change From Baseline in Hemoglobin, Total Protein, and Albumin at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: grams/deciliter (g/dL)
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
grams/deciliter (g/dL)
  Hemoglobin (HGB) | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Total Protein | -0.5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Albumin | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

9. Primary Outcome: Median Change From Baseline in Select Clinical Chemistry Parameters at Last Observation
Description: Includes median changes from baseline in total bilirubin, direct bilirubin, indirect bilirubin, blood urea nitrogen (BUN), creatinine, uric acid, calcium, magnesium, and glucose
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: milligrams/dL (mg/dL)
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
milligrams/dL (mg/dL)
  Total Bilirubin | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Direct Bilirubin | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Indirect Bilirubin | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Blood Urea Nitrogen (BUN) | -4.7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 5.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3.5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 3.8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -2.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Creatinine | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Uric Acid | -1.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Calcium | -0.2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Magnesium | -0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Glucose | -11 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 2 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 3 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -11 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

10. Primary Outcome: Median Change From Baseline in Sodium, Potassium, Chloride, and Bicarbonate at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: milliequivalents (mEq)/liter (L)
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
milliequivalents (mEq)/liter (L)
  Sodium | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Potassium | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Chloride | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Bicarbonate (venous) | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1.5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

11. Primary Outcome: Median Change From Baseline in Liver Function Tests at Last Observation
Description: Includes median changes in aspartate aminotransferase (AST), alanine aminotransferase (AST), gamma glutamyltransferase (GGT), and alkaline phosphatase
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: international units (IU)/L
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
international units (IU)/L
  Aminotransferase (AST) | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Alanine Aminotransferase (ALT) | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Gamma GT | -8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Alkaline Phosphatase | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 10 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

12. Primary Outcome: Median Change From Baseline in Thyroid-Stimulating Hormone (TSH) at Last Observation
Time Frame: Baseline, Last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: micro IU (mIU)/mL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
micro IU (mIU)/mL | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

13. Primary Outcome: Median Change From Baseline in Serum Creatine Kinase (CK), Amylase, and Lipase at Last Observation
Time Frame: Baseline, Last Observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: units (U)/L
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
units (U)/L
  Creatine Kinase (CK) | -17 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 21 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -43 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 13 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -11 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -16 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Amylase | 5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -12 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  Lipase | -1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 5 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 14 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -8 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 4 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

14. Primary Outcome: Median Change From Baseline in Free Triiodothyronine (T3) and Free Thyroxine (T4) at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication. Here "0" in the "overall number of participants analyzed" signifies that data not collected because none of the participants were evaluable for the specified arm.
Measure: Median (Full Range); unit: nanograms (ng)/dL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 0 | 6 | 0 | 0 | 20
nanograms (ng)/dL
  T3 (free) |  |  | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  |  | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.
  T4 (free) |  |  | -0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  |  | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

15. Primary Outcome: Median Change From Baseline in T4 at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: as for outcome 14
Measure: Median (Full Range); unit: micrograms (mcg)/dL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 8 | 8 | 20
micrograms (mcg)/dL | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.9 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -1.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.2 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.1 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

16. Primary Outcome: Median Change From Baseline in Urine WBC at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: as for outcome 14
Measure: Median (Full Range); unit: /high-powered field (HPF)
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 6 | 0 | 6 | 0 | 0 | 0 | 20
/high-powered field (HPF) |  | -1.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. |  |  |  | -1.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

17. Primary Outcome: Median Change From Baseline in Urine pH at Last Observation
Time Frame: Baseline, last observation (up to Day 85)
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: pH
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 20
pH | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.7 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.6 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | -0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.0 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan. | 0.3 [NA to NA] — Data for range was not collected, because analysis of median changes from baseline for laboratory parameters did not include range as part of the standard presentation per the statistical analysis plan.

18. Primary Outcome: Number of Participants With Abnormal and Clinically Relevant Changes in Blood Pressure
Description: Participants with maximum changes from baseline (defined as increases or decreases of greater than or equal to [≥]20 mmHg or ≥30 mmHg) in either standing or supine systolic blood pressure (SBP) or diastolic blood pressure (DBP) measured in millimeters mercury (mmHg).
Time Frame: Day 1 up to 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
Participants
  ≥30 mmHg decrease from baseline in supine SBP | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  ≥30 mmHg decrease from baseline in standing SBP | 3 | 0 | 0 | 0 | 1 | 3 | 1 | 4
  ≥20 mmHg decrease from baseline in supine DBP | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2
  ≥20 mmHg decrease from baseline in standing DBP | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3
  ≥30 mmHg increase from baseline in supine SBP | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  ≥30 mmHg increase from baseline in standing SBP | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 2
  ≥20 mmHg increase from baseline in supine DBP | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  ≥20 mmHg increase from baseline in standing DBP | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0

19. Primary Outcome: Number of Participants With Abnormal and Clinically Relevant Changes in Electrocardiogram (ECG) Parameters
Description: Participants with maximum changes from baseline (BSL) defined as: ≥25 to 50 percent (%) increase in maximum PR interval or QRS complex; increase from BSL of ≥30 milliseconds (msec) but <60 msec in corrected QT (QTc) interval or QTcF interval (QTc interval corrected using Fridericia's correction); or increase from BSL ≥60 msec in either QTc interval or QTcF interval.
Time Frame: Day 1 up to 85
Population: Safety Analysis Set: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
participants
  ≥25/50% increase from BSL in PR interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ≥25/50% increase from BSL in QRS complex | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ≥30 to <60 msec increase from BSL in QTc interval | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ≥60 msec increase from BSL in QTc interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ≥30 to <60 msec increase from BSL in QTcF interval | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  ≥60 msec increase from BSL in QTcF interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

20. Primary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) by Study Visit
Time Frame: Days -1, 8, 15, 29, 43, 57, and 85
Population: Safety Analysis Population
Measure: Number; unit: Participants
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8
Participants
  Day -1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 15 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Day 29 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 43 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 57 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 85 | 1 | 1 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 prior to infusion, 1, 2, 4, 8 and 12 hours and anytime on Days 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85 post-infusion
Population: Pharmacokinetic (PK) Parameter Analysis Set: All enrolled participants treated who had at least 1 of the PK parameters of interest. Here, "overall number of participants analyzed"= number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8
mcg*h/mL | 1175 (197.79) | 7588 (1297.1) | 86360 (12846) | 348800 (43230) | 33960 (4326.5) | 171100 (12762) | 269600 (27289)

22. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: as for outcome 21
Population: PK Parameter Analysis Set: All enrolled participants treated who had at least 1 of the PK parameters of interest. Here, "overall number of participants analyzed"= number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8
mcg/mL | 9.580 (0.69545) | 29.20 (4.3353) | 205.8 (29.743) | 687.3 (69.032) | 92.05 (27.124) | 409.6 (56.592) | 549.4 (60.738)

23. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8
hours | 1.49 [1.00 to 4.00] | 2.05 [2.00 to 4.00] | 2.00 [1.12 to 4.00] | 2.00 [1.02 to 8.00] | 1.56 [1.08 to 72.0] | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 4.03]

24. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: mL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 2 | 8 | 8 | 3
mL | NA (NA) — Vss could not be calculated for the 0.3 mg/kg dose since as per plan, reporting criteria for t1/2 were not met. The mean t1/2 could not be determined for the 0.3 mg/kg dose as the duration of sampling relative to the projected t1/2 was too short. | 3817 (601.08) | 3511 (517.52) | NA (NA) — Summary statistics were not calculated if fewer than 3 participants had reportable parameter values, as pre-specified. | 3822 (657.59) | 3782 (703.64) | 4063 (291.03)

25. Secondary Outcome: Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 21
Population: PK Parameter Analysis Set: All enrolled participants treated who had at least 1 of the PK parameters of interest. Here, "overall number of participants analyzed"= number of participants evaluable for this outcome measure and "0" in the "overall number of participants analyzed" signifies that data not collected because none of the participants were evaluable for the specified arm.
Measure: Geometric Mean (Standard Deviation); unit: mL/hr
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 0 | 6 | 6 | 0 | 8 | 8 | 3
mL/hr |  | 7.647 (1.9804) | 4.011 (0.72503) |  | 5.729 (1.2399) | 4.248 (0.77445) | 3.587 (0.32146)

26. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 2 | 8 | 8 | 3
hours | NA (NA) — The mean t1/2 could not be determined for the 0.3 mg/kg dose range as the duration of sampling relative to the projected t1/2 was too short. | 358.7 (50.603) | 637.8 (110.06) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. | 486.9 (92.644) | 657.5 (88.686) | 829.0 (82.286)

27. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)]
Description: AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf).
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 2 | 8 | 8 | 3
mcg*h/mL | NA (NA) — AUC(0-inf) could not be calculated for the 0.3 mg/kg dose since reporting criteria for t1/2 were not met. The mean t1/2 could not be determined for the 0.3 mg/kg dose range as the duration of sampling relative to the projected t1/2 was too short. | 8655 (1390.4) | 97010 (18085) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. | 36270 (5387.0) | 192600 (13512) | 323800 (34395)

28. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. Based on internal clinical pharmacology guidance on the most appropriate parameter calculations for this study design, data for Vz/F was not collected instead Vss was reported.
Time Frame: as for outcome 21
Population: Based on internal clinical pharmacology guidance on the most appropriate parameter calculations for this study design, Vz/F was not reported. Instead, Vss was reported.
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Percentage Change From Baseline in Total Dickkopf-1 (DKK-1) Concentrations Over Time
Time Frame: Day -1, Day 1 (predose and at end of infusion) and at 2, 4, 8, and 12 hours postdose, and Days 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57, and 85
Population: Pharmacodynamic (PD) Analysis Population: all enrolled participants who received at least 1 dose of study medication and had at least 1 PD parameter in at least 1 treatment period. Analytical qualification of a total DKK-1 assay was unsuccessful, thus no data was collected and reported.
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Mean Percentage Change From Baseline in Serum Procollagen Type 1 Amino-Terminal Propeptide (PINP) (ng/mL) Over Time
Description: Baseline calculated as average of Day -1 and Day 1 prior to infusion of PF-04840082
Time Frame: Baseline (Days -1, 1), Days 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85
Population: Pharmacodynamic (PD) Analysis Population: all enrolled participants who received at least 1 dose of study medication and had at least 1 PD parameter in at least 1 treatment period; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change from baseline
  Day 2 | 0.161 (6.9455) | 2.836 (6.4467) | 11.237 (16.8782) | 5.894 (10.8227) | 2.366 (5.9293) | 2.238 (9.8233) | -1.626 (11.2516) | 3.005 (6.4941)
  Day 3 | 7.908 (10.3904) | 3.745 (8.0952) | 10.157 (11.1075) | 8.461 (13.9663) | 10.031 (9.2134) | 11.711 (18.7964) | -3.213 (18.3073) | 4.963 (8.9468)
  Day 4 | 2.361 (16.5524) | -2.066 (6.7705) | 13.967 (17.9202) | 4.075 (5.5816) | 5.244 (8.4819) | 3.903 (11.3291) | -9.057 (18.0136) | -4.193 (9.1093)
  Day 5 | 8.794 (15.6171) | -2.352 (10.5552) | 7.884 (26.1801) | 5.535 (9.2328) | 12.242 (14.1055) | 5.619 (12.2245) | -12.708 (17.0940) | -3.344 (12.6299)
  Day 8 | 12.199 (20.7265) | 10.321 (10.8772) | 21.394 (20.6158) | 0.617 (8.3882) | 10.897 (20.3196) | 7.777 (16.0762) | 6.055 (12.4378) | -0.979 (9.7628)
  Day 15 | 8.524 (8.3551) | 7.618 (17.3215) | 28.710 (33.2390) | 12.031 (14.0186) | 9.904 (13.0457) | 15.259 (12.3700) | 9.717 (18.5300) | -0.968 (14.1064)
  Day 22 | 5.155 (14.1736) | 12.822 (9.7902) | 36.693 (29.1840) | 13.739 (13.9117) | 24.114 (20.7782) | 11.211 (13.9796) | 11.284 (13.1751) | -0.132 (9.1245)
  Day 29 | 2.579 (16.2957) | 5.117 (9.1142) | 23.742 (18.7153) | 16.135 (13.1185) | 26.118 (22.8948) | 12.405 (15.4178) | 10.753 (16.1139) | -6.509 (24.9432)
  Day 36 | -3.344 (17.0168) | 13.737 (10.2997) | 32.558 (50.4404) | 7.649 (18.2140) | 25.180 (18.4425) | 7.855 (11.6990) | 13.370 (17.6498) | 1.941 (12.6475)
  Day 43 | -1.986 (15.4137) | -17.799 (44.2793) | 19.420 (42.2273) | 0.720 (9.3270) | 28.914 (27.3598) | 10.576 (15.4128) | 12.696 (19.6629) | 1.210 (17.0653)
  Day 57 | 0.105 (26.5164) | 5.225 (14.3348) | 27.459 (60.2028) | -6.992 (20.6680) | 23.830 (28.0126) | 3.594 (23.5914) | 4.568 (21.1743) | -2.427 (12.3301)
  Day 85 | -7.489 (9.5892) | -4.566 (5.8947) | 37.825 (35.2720) | 5.423 (17.8942) | 22.304 (29.7686) | 1.623 (19.8165) | -2.263 (22.4866) | 0.820 (14.4801)

31. Secondary Outcome: Mean Percentage Change From Baseline in Serum n-Terminal Telopeptide(NTX) Over Time
Description: Baseline calculated as average of Day -1 and Day 1 prior to infusion of PF-04840082
Time Frame: Days -1, 1 (predose), 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85
Population: PD Analysis Population; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change from baseline
  Day 2 | -4.602 (14.2023) | -6.789 (9.8119) | -1.247 (19.0705) | 19.637 (13.9540) | -3.399 (21.0488) | -4.220 (39.6859) | -1.659 (19.1445) | -7.860 (16.6291)
  Day 3 | -17.167 (5.7802) | -1.748 (13.3302) | 2.418 (31.5323) | 13.956 (19.3949) | 0.893 (28.3001) | 4.121 (20.9339) | 18.209 (38.3564) | -4.200 (29.1776)
  Day 4 | -9.634 (9.5923) | 4.448 (18.3997) | 7.293 (24.6717) | 15.841 (23.4485) | 2.337 (24.1029) | -0.774 (42.0609) | 13.921 (27.0459) | 4.847 (22.2872)
  Day 5 | 2.826 (11.4062) | 8.577 (13.4307) | 18.005 (18.1277) | 17.300 (28.7024) | 5.471 (6.9326) | -2.630 (42.6402) | 0.658 (22.0426) | 7.604 (18.3770)
  Day 8 | 5.301 (9.8120) | 8.608 (11.9505) | 6.474 (20.9251) | 25.846 (41.5938) | 3.453 (23.3280) | 16.222 (23.3731) | -7.186 (12.9910) | 5.801 (19.8534)
  Day 15 | -7.765 (4.8847) | -11.284 (10.8652) | -1.807 (13.4761) | 10.608 (17.0266) | -13.589 (37.8165) | -1.536 (27.2663) | -17.954 (36.9722) | -11.942 (13.2393)
  Day 22 | -0.445 (22.3404) | 15.509 (33.1029) | 6.389 (13.9819) | 18.665 (28.1286) | 11.789 (26.3816) | 1.645 (27.2237) | -3.770 (12.9370) | 7.018 (36.6005)
  Day 29 | -0.026 (19.4086) | -4.254 (17.2335) | 17.712 (10.5885) | 33.244 (19.9530) | 7.721 (39.3020) | 11.095 (32.3792) | 0.979 (26.2735) | 5.779 (27.5110)
  Day 36 | -3.067 (17.7754) | 3.234 (24.2622) | 12.494 (12.9419) | 3.576 (15.1739) | 26.179 (24.2615) | 8.340 (33.1330) | -3.981 (20.5915) | 6.048 (31.9348)
  Day 43 | -7.690 (21.3058) | -3.596 (12.5937) | 0.833 (16.6770) | 14.111 (23.1987) | 25.679 (36.1569) | 13.512 (32.4953) | -1.915 (20.7555) | 0.609 (20.9022)
  Day 57 | 2.287 (20.6325) | 9.131 (14.1892) | 12.259 (18.8943) | 20.932 (22.0040) | 25.024 (33.4126) | 20.849 (62.3389) | -25.654 (35.7350) | -0.175 (24.4156)
  Day 85 | 5.677 (6.5738) | 14.354 (33.2027) | -3.162 (56.6723) | 20.327 (24.8686) | 12.477 (31.9743) | 7.108 (37.6896) | -5.121 (13.1626) | 1.615 (20.9010)

32. Secondary Outcome: Mean Percentage Change From Baseline in Serum Carboxy (C) Terminal Telopeptide (CTX) Over Time
Description: Baseline calculated as average of Day -1 and Day 1 prior to infusion of PF-04840082
Time Frame: Days -1, 1 (predose), 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85
Population: PD Analysis Population; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change
  Day 2 | 3.467 (7.6528) | 6.218 (19.6492) | 26.444 (16.5991) | 9.644 (6.9192) | 0.024 (14.1443) | 4.756 (16.3268) | 7.585 (8.7674) | 2.372 (27.8091)
  Day 3 | -4.472 (7.9083) | 4.296 (15.1105) | 16.416 (6.2517) | 11.628 (9.2015) | -0.980 (17.3430) | 6.211 (24.1040) | 14.878 (17.6179) | 9.334 (15.7981)
  Day 4 | -10.411 (13.5145) | 1.482 (14.9042) | 15.999 (18.0461) | -0.529 (14.2914) | -5.354 (25.1017) | -14.378 (12.3489) | 3.407 (20.9937) | 7.499 (15.6537)
  Day 5 | -8.039 (9.8536) | 8.380 (20.4009) | 9.864 (20.1860) | -0.322 (8.0655) | 0.462 (27.4688) | -6.551 (16.7397) | 11.802 (25.1567) | 3.983 (20.4928)
  Day 8 | -9.424 (10.3618) | -8.866 (19.8682) | 8.572 (24.7327) | -6.834 (9.6209) | -8.233 (31.2067) | -5.499 (21.6249) | -6.296 (17.1832) | 1.488 (15.6940)
  Day 15 | -12.864 (9.2562) | -7.907 (8.5077) | 24.010 (20.2593) | -2.931 (10.3678) | -12.009 (14.0871) | -4.800 (14.0773) | -4.586 (19.8401) | 7.668 (19.2344)
  Day 22 | -9.972 (14.6179) | -8.980 (16.1776) | 25.799 (20.0022) | -17.477 (9.9364) | -10.414 (10.1372) | -12.078 (17.7073) | -4.843 (14.4791) | 12.395 (42.6940)
  Day 29 | -6.741 (8.4135) | -11.367 (8.0673) | 27.694 (23.7259) | 1.130 (15.5004) | -19.376 (15.1382) | -3.761 (17.8403) | -5.356 (22.7410) | 2.626 (16.7445)
  Day 36 | 4.934 (19.2980) | -14.092 (14.6006) | 26.589 (18.1507) | -9.145 (22.6658) | -13.549 (16.1342) | -6.819 (30.2060) | 2.090 (15.8885) | 1.337 (21.1947)
  Day 43 | -9.903 (18.8829) | 0.422 (11.8856) | 18.554 (33.9325) | -8.871 (19.2661) | -1.681 (19.1395) | -8.608 (17.6558) | 5.776 (12.9204) | 1.531 (14.7672)
  Day 57 | 1.090 (16.2461) | -1.360 (11.7081) | 13.993 (17.1176) | -13.721 (13.0090) | 3.519 (29.4764) | -7.134 (28.0770) | -10.254 (16.1050) | 2.932 (23.9281)
  Day 85 | -5.989 (16.6472) | -5.584 (19.4223) | 33.724 (44.0981) | -14.097 (18.5865) | -4.368 (22.8715) | -12.647 (15.1312) | -9.104 (18.4964) | 2.521 (18.3823)

33. Secondary Outcome: Mean Percentage Change From Baseline in Serum Bone-Specific Alkaline Phosphatase (BSAP) Over Time
Description: Baseline calculated as average of Day -1 and Day 1 prior to infusion of PF-04840082
Time Frame: Days -1, 1 (predose), 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85
Population: PD Analysis Population; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change
  Day 2 | -6.185 (6.3059) | -2.849 (3.8567) | -0.796 (7.4823) | -7.570 (9.2328) | -0.796 (3.6143) | -6.334 (7.9459) | -3.927 (5.4622) | -3.934 (7.4244)
  Day 3 | -4.280 (9.5383) | 0.331 (6.4424) | 4.848 (10.6591) | 0.125 (7.8541) | 0.160 (7.3513) | -7.289 (5.5333) | -4.873 (14.7151) | -3.010 (8.1557)
  Day 4 | 0.929 (8.4449) | 0.729 (5.9355) | 5.189 (8.7365) | 2.074 (9.4077) | 2.460 (5.9179) | 0.052 (6.5211) | -2.325 (16.0997) | -0.876 (7.4064)
  Day 5 | 1.621 (11.3210) | 2.592 (6.4759) | 1.767 (8.0676) | 0.313 (3.9781) | 0.038 (5.5704) | -2.158 (10.6419) | -4.115 (16.0237) | -0.124 (10.4404)
  Day 8 | 6.038 (4.8726) | 7.438 (7.8948) | 6.823 (9.1449) | 5.260 (9.7094) | 0.558 (8.7457) | 2.468 (12.5723) | -0.332 (13.5092) | -0.594 (10.8209)
  Day 15 | 11.455 (7.6760) | 6.526 (6.5755) | 6.179 (9.1027) | 10.983 (10.9069) | 3.291 (9.4929) | 4.573 (9.0742) | 0.048 (8.8057) | -5.780 (12.2364)
  Day 22 | 19.200 (6.8095) | 15.884 (17.1866) | 4.513 (12.9814) | 9.570 (11.1603) | 3.469 (15.0685) | -2.533 (7.4853) | 2.937 (13.2892) | -2.589 (14.3755)
  Day 29 | 17.180 (7.2047) | 17.688 (18.6277) | 4.684 (14.0010) | 13.649 (7.9592) | -1.368 (16.3976) | -0.313 (14.4515) | 3.230 (16.5615) | -4.472 (15.3127)
  Day 36 | 12.815 (7.1986) | 10.798 (16.4632) | 9.205 (15.8163) | 9.652 (6.5596) | 7.952 (10.8748) | -0.917 (14.9214) | 1.002 (12.9844) | -0.863 (13.2753)
  Day 43 | 3.622 (5.8263) | 11.610 (14.5871) | 10.813 (12.7424) | 9.018 (8.0671) | 8.902 (16.7039) | 0.731 (11.6516) | 5.795 (15.4580) | 0.977 (13.0563)
  Day 57 | 6.766 (4.2535) | 0.848 (15.5889) | 7.169 (19.2122) | 0.851 (18.5419) | 9.197 (19.9274) | -10.431 (14.3542) | 0.676 (16.3864) | 0.155 (11.9164)
  Day 85 | 8.418 (9.2449) | -0.234 (8.3530) | 7.156 (8.6010) | 8.344 (5.4401) | 13.720 (17.5660) | -5.825 (16.8764) | 7.332 (12.0581) | 3.076 (13.2167)

34. Secondary Outcome: Mean Percentage Change From Baseline in Serum Osteocalcin Over Time
Description: Baseline calculated as average of Day -1 and Day 1 prior to infusion of PF-04840082
Time Frame: Days -1, 1 (predose), 2, 3, 4, 5, 8, 15, 22, 29, 36, 43, 57 and 85
Population: PD Analysis Population; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change
  Day 2 | 5.734 (14.0949) | 1.688 (11.1780) | 4.798 (8.2785) | 0.635 (10.1481) | 0.663 (8.3158) | -3.061 (12.9637) | -10.946 (16.5586) | 1.936 (9.1701)
  Day 3 | 4.252 (5.9602) | -2.471 (10.0364) | 3.026 (6.6556) | -0.209 (5.4522) | 3.157 (6.2435) | -3.711 (9.1520) | -7.423 (21.8432) | 3.742 (8.6378)
  Day 4 | 4.801 (15.6593) | 2.092 (13.5746) | 10.000 (11.8129) | 0.230 (8.3494) | 3.189 (12.2261) | -3.261 (14.2519) | -0.178 (14.0562) | 2.626 (9.7866)
  Day 5 | 6.641 (18.8735) | 4.175 (9.7966) | 1.586 (10.7697) | 7.592 (12.0591) | 6.756 (6.3289) | -0.848 (16.4937) | -3.098 (11.1147) | 1.747 (9.4714)
  Day 8 | 8.822 (22.5890) | 2.271 (9.4185) | 11.110 (6.1704) | -2.724 (8.4175) | -1.473 (7.9618) | 4.143 (16.5179) | 2.020 (8.1968) | 0.468 (9.2202)
  Day 15 | 4.055 (17.6355) | 3.056 (15.1080) | 12.216 (14.1642) | 1.975 (15.1871) | 4.501 (7.0609) | 3.062 (10.4890) | 0.989 (10.4834) | 3.223 (10.0156)
  Day 22 | 13.219 (12.8986) | 5.755 (8.6481) | 29.785 (19.5030) | 4.503 (9.3465) | 5.338 (7.8661) | 3.025 (11.8149) | 1.945 (5.9013) | 5.407 (9.6448)
  Day 29 | 11.576 (9.6497) | 5.871 (10.3258) | 18.627 (11.5843) | 10.099 (10.8958) | 1.437 (6.4453) | 9.743 (16.1027) | 2.127 (8.3314) | 3.921 (12.1504)
  Day 36 | 14.208 (21.3667) | 9.358 (5.7878) | 20.845 (19.4756) | 6.917 (16.2552) | 2.365 (5.0844) | 8.089 (14.6337) | 4.071 (8.5288) | 1.356 (13.0154)
  Day 43 | 6.087 (10.9388) | 8.222 (8.0005) | 8.185 (13.8026) | 3.429 (12.8258) | 8.281 (12.6603) | 7.902 (9.1879) | 4.218 (6.6123) | 1.908 (17.3185)
  Day 57 | 6.934 (12.8116) | 5.128 (10.0036) | 15.296 (36.6778) | -9.431 (15.5609) | 7.814 (19.6299) | 12.055 (27.4156) | -0.711 (11.7627) | 1.672 (12.3701)
  Day 85 | 5.766 (12.8626) | -7.261 (8.1118) | 30.350 (24.3439) | 6.667 (15.6370) | 2.338 (18.2941) | 0.554 (12.1071) | -2.414 (17.1454) | 1.329 (14.3518)

35. Secondary Outcome: Mean Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Day 85
Time Frame: Days -1 and 85
Population: PD Analysis Population; number analyzed=number of participants with an observation at the specified timepoints.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 20
percentage change
  AP Spine L1 BMD | -4.096 (7.5769) | 3.820 (2.8253) | -0.725 (2.8558) | -1.377 (6.5000) | 0.437 (6.1468) | -0.305 (4.2402) | -1.033 (3.4547) | -0.439 (3.7668)
  AP Spine L2 BMD | -1.441 (6.4764) | -0.816 (5.8942) | 0.454 (1.6845) | -0.200 (8.7398) | -0.940 (2.1560) | -0.890 (5.0854) | 0.609 (3.8245) | 1.060 (3.9478)
  AP Spine L3 BMD | 1.467 (5.3680) | -1.172 (6.4637) | 0.237 (3.0146) | -3.332 (4.5817) | 0.942 (2.8890) | 0.973 (5.3894) | 0.793 (4.8739) | -1.330 (3.1723)
  AP Spine L4 BMD | -1.908 (4.7541) | 2.443 (6.4076) | -1.553 (3.7424) | 1.228 (7.7207) | -0.171 (3.6823) | 0.470 (5.2763) | 0.171 (3.7706) | -1.288 (3.6274)
  AP Spine Total L1-L4 BMD | -1.356 (3.3947) | 0.975 (4.5713) | -0.914 (2.2948) | -0.918 (5.8689) | 0.144 (2.1232) | 0.095 (3.4250) | 0.206 (3.2457) | -0.794 (2.2182)

36. Secondary Outcome: Femoral Neck BMD at Day 85
Description: BMD was evaluated by dual energy X-ray absorptiometry (DXA).
Time Frame: Day 85
Population: PD Analysis Population. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Gram per centimeter square
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8 | 8 | 8 | 18
Gram per centimeter square | 0.7308 (0.09688) | 0.8357 (0.09877) | 0.8135 (0.10100) | 0.7954 (0.10295) | 0.8666 (0.11867) | 0.7185 (0.07402) | 0.8993 (0.06102) | 0.8362 (0.11301)

37. Secondary Outcome: Femoral Neck T-Score at Day 85
Description: BMD was evaluated by DXA. T-score was calculated based on actual measured bone density value and is the standardized scores that reflect the standard deviations (SDs) above/below the mean. A BMD T-score of -1.0 or more indicates normal bone density. T-score between -1.0 and -2.5 indicates low bone density known as osteopenia. A T-score of -2.5 or less is diagnostic of osteoporosis.
Time Frame: Day 85
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8 | 8 | 8 | 18
T-score | -1.2833 (0.81833) | -0.7333 (1.55906) | -1.2833 (0.36009) | -1.7600 (0.70922) | -0.9324 (1.14262) | -1.6500 (0.74066) | -0.8466 (0.73385) | -1.2278 (0.57477)

38. Secondary Outcome: Mean Percentage Change From Baseline in Distal Radius BMD at Day 85
Description: BMD was evaluated by DXA.
Time Frame: Baseline (Day -1), Day 85
Population: PD Analysis Population; Here, Overall number of participants analyzed=number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 8 | 8 | 7 | 17
percentage change
  Radius BMD | -0.138 (3.3241) | 1.673 (5.2845) | -1.545 (3.8933) | 1.226 (2.5319) | 1.387 (3.3849) | -1.223 (4.6806) | 6.485 (7.5097) | -0.610 (6.6493)
  Ulna BMD | -1.014 (4.1485) | 2.767 (6.7007) | -0.760 (2.0682) | 3.131 (2.8903) | 1.207 (3.0197) | -2.595 (2.6200) | 7.542 (7.5636) | -1.101 (7.2397)
  Forearm Total BMD | -8.608 (19.6096) | 0.716 (6.9188) | -1.253 (3.0603) | 7.744 (13.4882) | -0.823 (7.7854) | -2.087 (2.1496) | 6.944 (6.4528) | 2.439 (12.9063)

39. Secondary Outcome: PK/PD Model Describing the Relationship Between PF-04840082 PK Parameter Estimates/Concentrations and Changes in PD Endpoints
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 to Day 85
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04840082 0.3 mg/kg | PF-04840082 1.0 mg/kg | PF-04840082 6.0 mg/kg | PF-04840082 24.0 mg/kg | PF-04840082 3.0 mg/kg | PF-04840082 12.0 mg/kg | PF-04840082 18.0 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 1/8 | 0/8 | 1/20
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 6/6 | 5/6 | 5/8 | 6/8 | 6/8 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04840082 0.3 mg/kg (N=6) | PF-04840082 1.0 mg/kg (N=6) | PF-04840082 6.0 mg/kg (N=6) | PF-04840082 24.0 mg/kg (N=6) | PF-04840082 3.0 mg/kg (N=8) | PF-04840082 12.0 mg/kg (N=8) | PF-04840082 18.0 mg/kg (N=8) | Placebo (N=20)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04840082 0.3 mg/kg (N=6) | PF-04840082 1.0 mg/kg (N=6) | PF-04840082 6.0 mg/kg (N=6) | PF-04840082 24.0 mg/kg (N=6) | PF-04840082 3.0 mg/kg (N=8) | PF-04840082 12.0 mg/kg (N=8) | PF-04840082 18.0 mg/kg (N=8) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 3 | 2 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.